CLINICAL TRIAL: NCT05538065
Title: Optimizing Electronic Health Record Prompts With Behavioral Economics to Improve Prescribing for Older Adults
Brief Title: NUDGE-EHR Replication Trial at Mass General Brigham
Acronym: NUDGE-EHR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Massachusetts General Hospital (Other); National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Niteesh K. Choudhry, MD, PhD, Niteesh K. Choudhry, MD, PhD, Professor, Harvard Medical School, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2019A013684; R33AG057388 (NIH)
Record Dates: First submitted 2022-09-09; First posted 2022-09-13 (Actual); Results first posted 2025-04-01 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Aging; Benzodiazepine Sedative Adverse Reaction; Anticholinergic Adverse Reaction; Adverse Drug Event
Keywords: Benzodiazepine; Sedative hypnotic; Overprescribing; Anticholinergic
MeSH Terms: conditions — Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- No Alert (Usual Care) (No Intervention): Providers randomized to usual care will receive no intervention.
- Open Encounter + Pre-commitment (Experimental): There will be an enhanced EHR alert, known as a Best Practice Advisory [BPA], which will appear on each provider's EHR screen. We will also test a two-staged pre-commitment BPA in which the providers are prompted to discuss risks of the high-risk medications and share a handout about risks with their patients.
  Interventions: Other: Pre-commitment; Other: Enhanced Alert
- Open Encounter + Follow-up booster (Experimental): There will be an enhanced EHR alert, known as a Best Practice Advisory [BPA], which will appear on each provider's EHR screen. We will add a boostering option in the enhanced BPA, which is a provider-directed option for a follow-up in-basket message sent 4 weeks after the BPA is triggered.
  Interventions: Other: Follow-up booster Alert; Other: Enhanced Alert

INTERVENTIONS:
Other: Follow-up booster Alert — Once the order entry or open encounter alert displays, the provider will have the option to schedule a follow-up message that will be sent 4 weeks after the alert is triggered
  Arms: Open Encounter + Follow-up booster
Other: Pre-commitment — A two-staged pre-commitment electronic health record alert will be used. In the 1st alert, the providers will be prompted to discuss risks of these high-risk medications and share a handout about the risks with their patients, at their own discretion. The second alert will be either an order entry or open encounter alert, depending on the arm the provider is assigned to.
  Arms: Open Encounter + Pre-commitment
Other: Enhanced Alert — An enhanced alert (known as a Best Practice Advisory [BPA]) will appear on the provider's electronic health record screen and will contain several standard components such as information about why the medication is dangerous for their patient and an order set that will allow providers to order a gradual dose taper for their patient, order alternative medications, place a referral to a behavioral health specialist, provide instructions on how to make lifestyle modifications to improve patient symptoms, and add patient instructions for how to gradually taper off benzodiazepines and sedative hypnotics, as applicable.
  Arms: Open Encounter + Follow-up booster; Open Encounter + Pre-commitment

SUMMARY:
Prescribing of potentially unsafe medications for older adults is extremely common; benzodiazepines and sedative hypnotics are, for example, key drug classes frequently implicated in adverse health consequences for vulnerable older adults, such as confusion or sedation, leading to hospitalizations, falls, and fractures. Fortunately, most of these consequences are preventable. Physicians' lack of awareness of alternatives, ambiguous practice guidelines, and perceived pressure from patients or caregivers are among the reasons why these drugs are used more than might be optimal. Reducing inappropriate use of these drugs may be achieved through decision support tools for providers that are embedded in electronic health record (EHR) systems. While EHR strategies are widely used to support the informational needs of providers, these tools have demonstrated only modest effectiveness at improving prescribing. The effectiveness of these tools could be enhanced by leveraging principles of behavioral economics and related sciences.

DETAILED DESCRIPTION:
This is a cluster randomized control trial (RCT) to evaluate whether newly designed EHR-based tools designed using behavioral principles reduce inappropriate prescribing and adverse outcomes among older adults. This study will be conducted in outpatient primary care practices at Mass General Brigham (MGB), specifically Massachusetts General Hospital. MGB has a fully functional EHR, EpicCare, that supports computerized ordering of medications. MGB is comprised of 150 outpatient practices with over 1,800 physicians.

In this trial, approximately 190 primary care providers at MGH will be randomized to receive usual care or an active intervention. Providers randomized to one of the 2 selected treatment arms will receive an EHR tool to guide their care of eligible patients. They will be followed for 12 months. Providers randomized to usual care will receive no newly-designed EHR tool. Providers will receive these EHR tools for their patients who meet the following criteria: 1) older adults (aged 65 years or more), and 2) who have been prescribed at least 90 pills of benzodiazepine or sedative hypnotic or have been prescribed at least one active orders of at least 90 pills of two different anticholinergics in the last 180 days.

ELIGIBILITY:
Inclusion Criteria:

* Primary care provider at Mass General Brigham

Providers will receive these EHR tools for their patients who meet the following criteria:

1. older adults (aged 65 years or more)
2. who have been prescribed at least 90 pills of benzodiazepine or sedative hypnotic in the last 180 days.

Outcomes will be measured on the patient level.

Exclusion Criteria:

* N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2022-11-10 (Actual); Primary Completion 2024-03-15 (Actual); Study Completion 2024-06-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Niteesh K Choudhry, MD, PhD, Principal Investigator — Brigham and Women's Hospital
Locations (1):
- Mass General Brigham, Boston, Massachusetts, United States

REFERENCES:
- [Derived] Lauffenburger JC, Sung M, Glynn RJ, Keller PA, Robertson T, Kim DH, Bhatkhande G, Jungo KT, Haff N, Hanken KE, Isaac T, Choudhry NK. Electronic Health Record Intervention and Deprescribing for Older Adults: A Randomized Clinical Trial. JAMA. 2026 Jan 29:e2526967. doi: 10.1001/jama.2025.26967. Online ahead of print. PMID 41609788

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Primary care providers were cluster-randomized to these arms based on data available from the electronic health record and were not recruited directly for the trial or evaluated for effectiveness outcomes. Patients were also not intervened upon nor directly enrolled into the study. As such, we received a waiver of informed consent for participation.
Pre-assignment Details: Primary care providers were identified from electronic health record data and cluster randomized to a study arm. Patients who sought care from these primary care providers were identified based on electronic health record data for analyses and are classified as the participants. Providers were not assessed for effectiveness outcomes.
Units Other Than Participants: Primary care providers
Period: Overall Study
Arm/Group | No Alert (Usual Care) | Open Encounter + Pre-commitment | Open Encounter + Follow-up Booster
Started | 396; 67 Primary care providers | 394; 67 Primary care providers | 356; 67 Primary care providers
Completed | 396; 67 Primary care providers | 394; 67 Primary care providers | 356; 67 Primary care providers
Not Completed | 0; 0 Primary care providers | 0; 0 Primary care providers | 0; 0 Primary care providers

BASELINE CHARACTERISTICS:
Population: All of these baseline measures are for the patients included in analyses in the data. Data from primary care providers (the unit of randomization) was not collected at baseline nor in follow-up.
Groups:
- Total: Total of all reporting groups
Arm/Group | No Alert (Usual Care) | Open Encounter + Pre-commitment | Open Encounter + Follow-up Booster | Total
Number analyzed (Participants) | 396 | 394 | 356 | 1146
Age, Continuous [Mean (Standard Deviation); unit: years] | 73.5 (6.4) | 73.7 (6.5) | 73.6 (6.5) | 73.6 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 275 | 276 | 248 | 799
  Male | 121 | 118 | 108 | 347
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 21 | 26 | 33 | 80
  Not Hispanic or Latino | 364 | 348 | 306 | 1018
  Unknown or Not Reported | 11 | 20 | 17 | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 2
  Asian | 12 | 11 | 13 | 36
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 1 | 1
  Black or African American | 12 | 14 | 10 | 36
  White | 350 | 347 | 298 | 995
  More than one race | 12 | 15 | 25 | 52
  Unknown or Not Reported | 10 | 6 | 8 | 24

OUTCOME MEASURES:

1. Primary Outcome: Change in Inappropriate Prescribing
Description: This outcome is measured as a composite of 1) discontinuation of study high-risk medications (i.e., active discontinuation or lack of an order during follow-up) or 2) ordering a dose taper (for benzodiazepine or sedative hypnotics) using EHR data by the primary care provider included in the study arm. If any of these actions occurred by the primary care provider, then the patient was considered to have had a change in prescribing (i.e., a reduction in inappropriate prescribing). This outcome was measured as a binary outcome.
Time Frame: Each patient was assessed beginning from the date in which they were identified as eligible (i.e., meeting the inclusion criteria) until the end of a 16-month follow-up; the outcome time frame varied by participant
Population: Patients who met eligibility criteria for inclusion in the analysis (adults ≥65 years, who were prescribed ≥90 pills of benzodiazepine, strongly anticholinergic medication, or sedative hypnotic in the last 180 days and had an office or telemedicine visit with a primary care provider who was assigned to a study arm), as measured from EHR system data.
Measure: Count of Participants; unit: Participants
Arm/Group | No Alert (Usual Care) | Open Encounter + Pre-commitment | Open Encounter + Follow-up Booster
Number analyzed (Participants) | 396 | 394 | 356
Participants | 106 | 145 | 122
Statistical Analysis 1: Comparison: No Alert (Usual Care) vs Open Encounter + Pre-commitment; Outcomes were evaluated using generalized estimating equations with a log link and binary errors, adjusting for provider-level clustering and Holm-Bonferroni multiple comparisons; Test type: Superiority; p = 0.002, Regression, Logistic — Adjusted for multiple comparisons; Risk Ratio (RR) = 1.40, 95% CI 2-sided [1.10 to 1.78]
Statistical Analysis 2: Comparison: No Alert (Usual Care) vs Open Encounter + Follow-up Booster; [analysis description as in outcome 1, analysis 1]; Test type: Superiority; p = 0.039, Regression, Logistic — Adjusted for multiple comparisons; Risk Ratio (RR) = 1.26, 95% CI 2-sided [1.01 to 1.57]

2. Secondary Outcome: Quantity of High-risk Medication Prescribed
Description: This outcome is measured on the patient level as the number of pills of high-risk medications prescribed to patients by providers over the follow-up, measured within the EHR system. This outcome was measured as a continuous outcome.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of pills
Arm/Group | No Alert (Usual Care) | Open Encounter + Pre-commitment | Open Encounter + Follow-up Booster
Number analyzed (Participants) | 396 | 394 | 356
Number of pills | 398.6 (439.4) | 422.5 (470.9) | 437.9 (481.6)
Statistical Analysis 1: Comparison: No Alert (Usual Care) vs Open Encounter + Pre-commitment; Outcomes were evaluated using generalized estimating equations with an identity link and normally-distributed errors, adjusting for provider-level clustering and Holm-Bonferroni multiple comparisons; Test type: Superiority; p = 0.386, Regression, Linear — Adjusted for multiple testing; Mean Difference (Final Values) = 29.0, 95% CI 2-sided [-36.6 to 94.6]
Statistical Analysis 2: Comparison: No Alert (Usual Care) vs Open Encounter + Follow-up Booster; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 272, Regression, Linear — Adjusted for multiple comparisons; Mean Difference (Final Values) = 38.1, 95% CI 2-sided [-29.9 to 106.1]

3. Secondary Outcome: Cumulative Lorazepam Milligram Equivalents Prescribed
Description: This outcome is measured on the patient level as the number of lorazepam milligram equivalents of benzodiazepine and sedative hypnotic ("Z-drug") prescribed to patients by providers over the follow-up, measured within the EHR system. This outcome was measured as a continuous outcome.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: lorazepam milligram equivalents
Arm/Group | No Alert (Usual Care) | Open Encounter + Pre-commitment | Open Encounter + Follow-up Booster
Number analyzed (Participants) | 396 | 394 | 356
lorazepam milligram equivalents | 238.7 (461.6) | 220.1 (413.9) | 259.7 (601.3)
Statistical Analysis 1: Comparison: No Alert (Usual Care) vs Open Encounter + Pre-commitment; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.657, Regression, Linear — Adjusted for multiple testing; Mean Difference (Final Values) = -13.8, 95% CI 2-sided [-74.5 to 47.0]
Statistical Analysis 2: Comparison: No Alert (Usual Care) vs Open Encounter + Follow-up Booster; [analysis description as in outcome 2, analysis 1]; Test type: Superiority; p = 0.696, Regression, Linear; Adjusted for multiple testing; Mean Difference (Final Values) = 15.1, 95% CI 2-sided [-60.7 to 91.0]

ADVERSE EVENTS:
Time Frame: 16 months
Description: Deaths and adverse events are reported for patients who were included in the analyses for the trial. Deaths and adverse events were not collected, monitored, or assessed for providers. For patients, we used an automatic adverse event reporting system to monitor for any AEs that occurred, which were routinely reviewed by quality and safety specialists at the institution. In addition, for patients, we retrospectively identified patient deaths through a retrospective review within the EHR.
Arm/Group | No Alert (Usual Care) | Open Encounter + Pre-commitment | Open Encounter + Follow-up Booster
All-Cause Mortality (participants affected / at risk) | 14/396 | 7/394 | 6/356
Serious Adverse Events (participants affected / at risk) | 0/396 | 0/394 | 0/356
Other Adverse Events (participants affected / at risk) | 0/396 | 0/394 | 0/356

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-04-14): https://cdn.clinicaltrials.gov/large-docs/65/NCT05538065/Prot_SAP_001.pdf